CLINICAL TRIAL: NCT03854539
Title: Salivary Alpha Amylase as a Biomarker of Transdermal Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Tech University (Other)
Responsible Party: Principal Investigator, Rodney Roosevelt, Assistant Professor, Arkansas Tech University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Roosevelt-1
Record Dates: First submitted 2018-04-19; First posted 2019-02-26 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: No Condition Salivary Alpha Amylase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Active Stimulation 0.5 (Experimental): 0.5 mA intermittent transdermal stimulation of the aurical vagus stimulation 30 seconds on/30 seconds off for five cycles
  Interventions: Other: Transdermal Vagus Nerve Stimulation
- Sham Stimulation (Sham Comparator): 0.5mA intermittent transdermal stimulation of the aurical vagus stimulation5 Hz 30 seconds on/30 seconds off for five cycles
  Interventions: Other: Transdermal Vagus Nerve Stimulation
- No Stimulation (No Intervention): 0.0 mA (sham) intermittent transdermal stimulation of the aurical vagus stimulation, 0 Hz 30 seconds on/30 seconds off for five cycles
- Active Stimulation 1.0 (Experimental): 0.5 mA intermittent transdermal stimulation of the aurical vagus stimulation 30 seconds on/30 seconds off for five cycles.
  Interventions: Other: Transdermal Vagus Nerve Stimulation
- Active Stimulation 0.25 (Experimental): 0.25 mA intermittent transdermal stimulation of the aurical vagus stimulation 30 seconds on/30 seconds off for five cycles
  Interventions: Other: Transdermal Vagus Nerve Stimulation

INTERVENTIONS:
Other: Transdermal Vagus Nerve Stimulation — intermittent transdermal stimulation of the aurical vagus
  Arms: Active Stimulation 0.25; Active Stimulation 0.5; Active Stimulation 1.0; Sham Stimulation

SUMMARY:
The proposed project tests the hypothesis that salivary alpha amylase concentration is a reliable biomarker of the effect of transdermal vagus nerve stimulation (tVNS) in humans.

DETAILED DESCRIPTION:
The study examines the capacity of tVNS to alter the concentrations of salivary alpha amylase. Changes in salivary alpha amylase concentrations reflect alteration of CNS structures anatomically linked to the vagus, thus alertation of alpha amylase would indicate the efficacy of tVNS. This study is intended to study basic mechanisms and is not directed toward the treatment of any disease state. Particapants taking part in the study will spend about one hour in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Alpha Amylase concentration. | Within single one hour session change in concentration immediately prior to and following stimulation and 5 minutes post-stimulation
  Biomarker of autonomic arousal level

SECONDARY OUTCOMES:
Change in Heart Rate Variability. | Within single one hour session change in heart rate variability immediately prior to and following stimulation period.
  Change in beat to beat interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Tech University, Russellville, Arkansas, United States